CLINICAL TRIAL: NCT06738277
Title: A Phase 1, Randomized, Open-label, 2-arm, Parallel Design Study in Normal Healthy Subjects to Evaluate Pharmacokinetics, Safety, and Tolerability of Bmab 1200 -Autoinjector (Biosimilar Ustekinumab) After Single Subcutaneous Injection in Comparison With Bmab 1200 -Prefilled Syringe (Biosimilar Ustekinumab)
Brief Title: This is Comparative Study in Normal Healthy Subjects to Evaluate Pharmacokinetics, Safety, Tolerability of Bmab 1200 -Autoinjector (AI) After Single Subcutaneous Injection (45 mg) in Comparison With Bmab 1200 -Prefilled Syringe (PFS).
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biocon Biologics UK Ltd (Industry)
Responsible Party: Sponsor
Organization: Biocon Limited (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIO-USTEKI-104
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Moderate to Severe Chronic Plaque Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bmab 1200 AI (Biosimilar Ustekinumab) (Experimental)
  Interventions: Drug: Bmab 1200 (Biosimilar Ustekinumab)
- Bmab 1200 PFS (Biosimilar Ustekinumab) (Active Comparator)
  Interventions: Drug: Bmab 1200 (Biosimilar Ustekinumab)

INTERVENTIONS:
Drug: Bmab 1200 (Biosimilar Ustekinumab) — Dosage Form: injection, Strength(s): 45 mg/ 0.5 mL Route of Administration: Subcutaneous Frequency and Dose: 45 mg, single dose

SUMMARY:
This is an open-label, 2-arm parallel-group study in normal healthy subjects to evaluate pharmacokinetics, safety, tolerability of Bmab 1200 -autoinjector (AI) after single subcutaneous injection (45 mg) in comparison with Bmab 1200 -prefilled syringe (PFS).

DETAILED DESCRIPTION:
Bmab 1200 is being developed as a proposed biosimilar product to the reference product Stelara® in accordance with EU and US biosimilar guidelines. The currently available Bmab 1200 formulation is administered via SC injection using PFS (similar to the reference product Stelara®). The main purpose of this study is to establish the PK equivalence of Bmab 1200 -AI following a single SC injection ( 45 mg) in comparison with Bmab 1200 -PFS. AI and PFS are self-injectable devices that can deliver drugs through the SC route. This study will also assess the safety and tolerability of Bmab 1200 AI in comparison with Bmab 1200 PFS. This will enable the licensure of AI to improve patient compliance through controlled and standardized administration of Bmab 1200

ELIGIBILITY:
Inclusion Criteria:

* a.Non-smokers, healthy, adult, human volunteers between 18 to 55 years of age (both inclusive).

  b.Having BMI between 18.5 to 28.0 m2 and having a body weight between 60 kg and 90 kg (both inclusive for both parameters).

  c.Not having any significant diseases or clinically significant abnormal findings during screening, medical history, clinical examination, laboratory evaluations, 12-lead ECG and X-ray chest (P/A view) recordings.

  d.Able to understand and comply with the study procedures, in the opinion of the investigator.

  e.Able to give voluntary written informed consent for participation in the study.

  f.Subjects should not receive a BCG vaccine within 1 year before dosing and agree to not take it during the study and at least 1 year after dosing.

  g.Subjects will agree not to receive live vaccination during the study. h.Subject will agree not to donate blood/ plasma/ platelets during the study and at least 3 months after the end of study.

  i.For male subjects i.Subjects agree to use effective contraception (e.g. Double barrier method) and refrain from donation of sperm from check-in until 90 days after the end of study.

  j.In case of female subjects: i.Surgically sterilized at least 6 months prior to study participation Or If subject is of child-bearing potential, is willing to use a suitable and effective double barrier contraceptive method or intrauterine device during the study and till 4 months after the end of study.

Or Post-menopausal women. And ii.Serum pregnancy test must be negative. iii.Subjects will agree to refrain from donation of ova from check-in until 90 days after the end of study.

Exclusion Criteria:

* a. Known hypersensitivity or idiosyncratic reaction to ustekinumab or any excipients or any related drug or any substance (specifically any biologic product or the constituents of Bmab 1200).

  b. Known hypersensitivity to host cell [ murine myeloma cell or Chinese hamster ovary cells] derived proteins, latex), food, or other substance.

  c. History or presence of any disease or condition which might compromise the haemopoietic, renal, hepatic, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal, or any other body system.

  d. Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes.

  e. Use or intend to use any prescription medications/products or other acceptable concomitant Medications within 30 days prior to dosing or slow-release medications/products considered to still be active within 14 days prior to check-in.

  f. Use or intend to use any nonprescription medications/ products, including vitamins, minerals, and phytotherapeutic/ herbal/ plant-derived preparations within 7 days prior to check-in.

  g. Use of any vaccine from 4 weeks prior to screening.

  h. The QTc interval more than 450 ms for male and more than 460 ms for female at the time of screening.

  i. Any history or presence of asthma (including aspirin-induced asthma) or nasal polyp or NSAIDs induced urticaria.

  j. A recent history of harmful use of alcohol (less than 2 years), or consumption of alcohol or alcoholic products within 48 hours prior to receiving study drug.

  k. Smokers, or who have smoked within the last six months prior to the start of the study.

  l. The presence of clinically significant abnormal laboratory values during screening.

  m. Use of any recreational drugs or history of drug addiction or testing positive in pre-study drug scans.

  n. History or presence of seizure or psychiatric disorders.

  o. A history of difficulty with donating blood.

  p. Donation of blood (1 unit or 350 mL) or plasma/ platelets in the last 90 days prior to screening until 3 months after the end of study visit.

  q. Participation in a clinical study involving the administration of an investigational drug in the past 90 days or 5 half-lives (whichever is longer), prior to dosing.

  r. A positive hepatitis screen including hepatitis B surface antigen and/or HCV antibodies.

  s. A positive test result for HIV antibody (I &/or 2).

  t. Current history of active infections, including significant localized infections, cough or fever, or current /previous history of recurrent or chronic infections. (At screening and within 1 week prior to study drug administration).

  u. History of active tuberculosis (TB) or presence of active or latent TB. A positive result for IGRA (Interferon Gamma Release Assay) test at screening.

  v. Known history of previous exposure to ustekinumab or ustekinumab biosimilar, or any IL-12 or IL-23 monoclonal antibodies, approved or investigational.

  w. Consumption of grapefruit or grapefruit products within 72 hours prior to dosing.

  x. An unusual diet, for whatever reason (for example, fasting, high potassium or low sodium), for four weeks prior to receiving the study medicine. In any such case, subject selection will be at the discretion of the Principal Investigator.

  y. Ingestion of poppy seed-containing foods or beverages within 7 days prior to check-in.

  z. Receipt of blood products within 2 months prior to check-in. aa. Poor peripheral venous access.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 186 (Actual)
Dates: Start 2025-01-09 (Actual); Primary Completion 2025-07-12 (Actual); Study Completion 2025-07-12 (Actual)

PRIMARY OUTCOMES:
Cmax | Week 16
  Maximum observed concentration (Cmax) of drug Bmab 1200
AUCo-∞ | Week 16
  Comparison of area under the concentration-time curve from time 0 to infinity (AUC0-inf)

SECONDARY OUTCOMES:
AUCo-t | Week 16
  Area Under the serum Concentration versus time curve from time 0 to the last sampling time at which concentrations were at or above the limit of quantification
Tmax | Week 16
  Time to maximum observed concentration
AUC_%Extrap_obs | Week 16
  % of the AUC that has been derived after extrapolation
ƛz | Week 16
  Elimination rate constant
Vd | Week 16
  Volume of distribution
Cl | Week 16
  drug clearance
t1/2 | Week 16
  Apparent terminal elimination half-life

CONTACTS AND LOCATIONS:
Locations (1):
- Lambda Therapeutic Research Ltd, Ahmedabad, India